CLINICAL TRIAL: NCT04470518
Title: Impact of a Diagnostic Algorithm on Antibiotic Prescribing Rate and Further Management of Acutely Ill Children Presenting to Ambulatory Care: Multicentre, Cluster-randomized, Parallel Group Pragmatic Trial
Brief Title: Impact of Clinical Guidance & Point-of-care CRP in Children: the ARON Project
Acronym: ARON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); University Ghent (Other); Universiteit Antwerpen (Other); University of Liege (Other); Vrije Universiteit Brussel (Other); Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Jan Verbakel, Professor Doctor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S62005
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Infection
Keywords: antibiotic prescription; infections; decision tree; point-of-care C-reactive protein test; safetynet advice
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: multicentre, cluster-randomized, parallel group pragmatic trial
Masking Description: Owing to study procedures, children, their parents and physicians will not be masked to the practices' random allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Diagnostic algorithm (Active Comparator): diagnostic algorithm including a standardised clinical assessment, a Point-of-care C-reactive protein test, and safety netting advice
  Interventions: Other: diagnostic algorithm
- Usual care (No Intervention): In the control arm, patients will receive 'usual care' left at the discretion of the treating physician.
  Apart from the general training session for all participating physicians they have attended prior to recruitment and randomization, physicians in the control arm will not receive additional tools.
  They are expected (but not forced) to follow the Belgian guidelines (as described in "BAPCOC National guidelines and the RIZIV consensus meeting "Rational use of antibiotics in children").

INTERVENTIONS:
Other: diagnostic algorithm — Guidance will be part of a diagnostic algorithm which includes clinically guided point-of-care C-reactive protein testing and safety netting advice to inform parents on what to expect and what to look out for. A selection of clinical features will be assessed and recorded by the physician in the patient's health record and on the e-CRF, including the clinical decision tree (clinician's gut feeling, body temperature, dyspnea).
  The safety-netting advice will be supported by a parent information booklet, based on previous research (the "When should I worry"-interactive booklet (a guide to Coughs, Colds, Earache & Sore Throats), the "Mijn kind heeft koorts" booklet (Eefje de Bont, www.thuisarts.nl), and the "Caring for children with coughs"-leaflet (information about how to look after a child who has a cough and when to see the doctor)).
  Arms: Intervention: Diagnostic algorithm

SUMMARY:
Impact of clinical guidance & point-of-care CRP test in children: the ARON project Trial Design: multicentre, cluster-randomized, parallel group pragmatic trial Trial Participants and setting: Children aged 6 months to 12 years of age with an acute illness episode presenting to in-hours general practice or out-of-hospital community paediatrics offices

Intervention(s) Diagnostic algorithm:

1. Clinical decision tree: clinician's gut feeling something is wrong, dyspnea, temperature ≥40ºC
2. YES to any : point-of-care CRP ≥5mg/L: additional testing or refer to secondary care <5mg/L: safety netting*, only prescribe antibiotics if advised (guidelines)
3. NO to all : are AB considered? YES : point-of-care CRP ≥5mg/L: safety netting*, only prescribe antibiotics if advised (guidelines) <5mg/L: safety netting*, do not prescribe antibiotics NO: safety netting

   *safety netting advice:
   * inform parents on what to expect and what to look out for
   * interactive parent information booklet based on previous research

   Control: Diagnosis and Treatment/Management as per usual care:

   - guidance on AB prescribing:

   o Belgische Commissie voor de Coördinatie van het Antibioticabeleid (BAPCOC) guide (updated November 2019)

   o RIZIV consensus meeting report "Antibiotics in children in ambulatory care"

   Primary Endpoint: Antibiotic prescribing rate at index consultation

   Secondary Endpoint(s)

   - time until full clinical recovery (during follow up (day 1 to day 30))

   - additional investigations (at index consultation and/or during follow up (day 1 to day 30))

   - re-consultation (during follow up (day 1 to day 30))

   - antibiotic prescribing rate (during follow up (day 1 to day 30))

   Exploratory endpoints at the index consultation:
   * additional investigations (X-Ray, blood tests, urine tests, etc.)

   During a follow-up period (day 1 to day 30):

   - referral to hospital

   - additional investigations (X-Ray, blood tests, urine tests, etc.)
   * patients with full clinical recovery at day 7 and day 30
   * admission to hospital
   * mortality
   * cost-effectiveness
   * patient satisfaction
   * qualitative study: endpoints

   Planned Sample Size: 7000 Timing of the intervention: Intervention at index consultation (at presentation to primary care) Follow-up duration: 30 days follow-up Duration of the trial (FPI-CSR): 43 months

DETAILED DESCRIPTION:
The investigators aim to strengthen the assessment of acutely ill children in primary care, by introducing a diagnostic algorithm that can decrease antibiotic prescribing.

In light of the prior evidence and its results so far, the ARON trial will test the impact of a diagnostic algorithm including a standardised clinical assessment, a POC CRP test, and safety netting advice.

Therefore, the investigators propose to assess the clinical and cost-effectiveness of a diagnostic algorithm which includes a decision tree, POC CRP and safety netting advice in acutely ill children aged 6 months to 12 years of age presenting to ambulatory care, on AB prescribing, referral/admission to hospital, additional testing, mortality, and patient satisfaction.

More specifically, the investigators' research question is whether this diagnostic algorithm is able to safely reduce antibiotic prescribing in acutely ill children presenting to ambulatory care.

The decision whether or not to conduct a POC CRP test will depend on the standardized clinical assessment, i.e. a validated clinical decision tree, and subsequently for low-risk children on the intention to prescribe AB.

The investigators will provide clear evidence-based guidance on how to interpret the CRP test result as outlined below.

A process evaluation will examine how clinicians use CRP testing in their practice and how parents experience these consultations.

The investigators propose a study, where children (6 months to 12 years of age) will be randomised to (a) a diagnostic algorithm with CRP testing and specific guidance on when to prescribe AB or (b) usual care. CRP testing will be done using a finger prick test (result within 4 minutes). The CRP level will then be given to the clinician who will communicate the result to the child/parents.

The investigators aim to recruit 7000 children and will collect data registered by the participating physician, from the child's health record and children/parents directly. The investigators will describe how the intervention has worked in practice and how clinicians/parents have experienced these consultations.

Guidance will be part of a diagnostic algorithm which includes clinically guided POC CRP testing and safety netting advice to inform parents on what to expect and what to look out for.

Individual interviews will be conducted with clinicians and parents taking part in the trial within 30 days after the first contact consultation, to explore the social processes influencing embedding of the intervention within practice, and behaviour change techniques.

These individual telephone interviews will be performed with a selection of parents to address whether their concerns were discussed appropriately and whether their expectations were met and how they experienced the consultation and/or POC CRP testing.

The safety-netting advice will be supported by a parent information booklet, based on previous research (the "When should I worry"-interactive booklet (a guide to Coughs, Colds, Earache & Sore Throats), the "Mijn kind heeft koorts" booklet (Eefje de Bont, www.thuisarts.nl), and the "Caring for children with coughs"-leaflet (information about how to look after a child who has a cough and when to see the doctor)).

The findings of this study could change the practice of ambulatory care physicians and might be of great interest to parents and childcare providers. The investigators will publish the findings of this research in academic journals, present at national conferences and discuss results with groups responsible for the national guidance on how to assess acutely ill children (Domus Medica, SSMG).

ELIGIBILITY:
Inclusion Criteria for practices:

* Being able to recruit acutely ill children (ideally consecutively)
* Agree to the terms of the clinical study agreement.

Exclusion Criteria for practices:

* Currently using a POC CRP device as part of their routine care
* No practices will be excluded on other grounds than the above. Age, demographics, geographic region will not be used to exclude eligible practices. This will provide us with a real-life, representative subset of ambulatory care physicians.

Inclusion criteria for children

* Children aged 6 months to 12 years, provided informed consent can be obtained
* presenting with an acute illness episode that started maximum 10 days before the index consultation

Exclusion criteria for children

* Children who were previously included in this trial
* children with an underlying known chronic condition (e.g. asthma, immune deficiency)
* clinically unstable warranting immediate care
* immunosuppressant medication taken in the previous 30 days
* trauma as the main presenting problem
* antibiotics taken in the previous 7 days
* Unwillingness or inability to provide informed consent

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6750 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Y Verbakel, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- GPs associated with KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data from this trial will not be published in the public domain. Deidentified participant data is available for further analyses. Requests for data, with justification, should be sent to Jan Verbakel (Jan . verbakel @ kuleuven.be, Tine De Burghgraeve (tine . deburghgraeve @ kuleuven.be. The trial protocol is available online for an indefinite period.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Study protocol is published and accessible. SAP, CSR, ICF and analytical code will be available after publishing the results in a medical journal. Individual patient data from this trial will not be published in the public domain.
Access Criteria: Individual patient data from this trial will not be published in the public domain. Deidentified participant data is available for further analyses. Requests for data, with justification, should be sent to JYV, TDB, or RB. The trial protocol is available online for an indefinite period.
URL: https://pubmed.ncbi.nlm.nih.gov/34980633/

REFERENCES:
- [Background] Verbakel JY, Lemiengre MB, De Burghgraeve T, De Sutter A, Aertgeerts B, Bullens DMA, Shinkins B, Van den Bruel A, Buntinx F. Point-of-care C reactive protein to identify serious infection in acutely ill children presenting to hospital: prospective cohort study. Arch Dis Child. 2018 May;103(5):420-426. doi: 10.1136/archdischild-2016-312384. Epub 2017 Dec 21. PMID 29269559
- [Background] Verbakel JY, Aertgeerts B, Lemiengre M, Sutter AD, Bullens DM, Buntinx F. Analytical accuracy and user-friendliness of the Afinion point-of-care CRP test. J Clin Pathol. 2014 Jan;67(1):83-6. doi: 10.1136/jclinpath-2013-201654. Epub 2013 Sep 11. No abstract available. PMID 24025452
- [Background] Verbakel JY, Lemiengre MB, De Burghgraeve T, De Sutter A, Aertgeerts B, Shinkins B, Perera R, Mant D, Van den Bruel A, Buntinx F. Should all acutely ill children in primary care be tested with point-of-care CRP: a cluster randomised trial. BMC Med. 2016 Oct 6;14(1):131. doi: 10.1186/s12916-016-0679-2. PMID 27716201
- [Derived] Verbakel JY, Burvenich R, D'hulster E, De Rop L, Van den Bruel A, Anthierens S, Coenen S, De Sutter A, Heytens S, Joly L, Digregorio M, Laenen A, Luyten J, De Burghgraeve T. A clinical decision tool including a decision tree, point-of-care testing of CRP, and safety-netting advice to guide antibiotic prescribing in acutely ill children in primary care in Belgium (ARON): a pragmatic, cluster-randomised, controlled trial. Lancet. 2025 Oct 11;406(10512):1599-1610. doi: 10.1016/S0140-6736(25)01239-5. Epub 2025 Sep 25. PMID 41016406
- [Derived] Verbakel JYJ, De Burghgraeve T, Van den Bruel A, Coenen S, Anthierens S, Joly L, Laenen A, Luyten J, De Sutter A. Antibiotic prescribing rate after optimal near-patient C-reactive protein testing in acutely ill children presenting to ambulatory care (ARON project): protocol for a cluster-randomized pragmatic trial. BMJ Open. 2022 Jan 3;12(1):e058912. doi: 10.1136/bmjopen-2021-058912. PMID 34980633

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: general practices
Groups:
- Intervention: Diagnostic Algorithm: diagnostic algorithm including a standardised clinical assessment, a Point-of-care C-reactive protein test, and safety netting advice
  diagnostic algorithm: Guidance will be part of a diagnostic algorithm which includes clinically guided point-of-care C-reactive protein testing and safety netting advice to inform parents on what to expect and what to look out for. A selection of clinical features will be assessed and recorded by the physician in the patient's health record and on the e-CRF, including the clinical decision tree (clinician's gut feeling, body temperature, dyspnea).
  The safety-netting advice will be supported by a parent information booklet, based on previous research (the "When should I worry"-interactive booklet (a guide to Coughs, Colds, Earache & Sore Throats), the "Mijn kind heeft koorts" booklet (Eefje de Bont, www.thuisarts.nl), and the "Caring for children with coughs"-leaflet (information about how to look after a child who has a cough and when to see the doctor)).
Period: Overall Study
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Started | 2988; 82 general practices | 3762; 89 general practices
Completed | 2988; 82 general practices | 3762; 89 general practices
Not Completed | 0; 0 general practices | 0; 0 general practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care | Total
Number analyzed (Participants) | 2988 | 3762 | 6750
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.7 [1.6 to 7.1] | 3.9 [1.8 to 7.2] | 3.75 [1.75 to 7.08]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  boy | 1566 | 1881 | 3447
  girl | 1421 | 1881 | 3302
  prefer not to say | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 2988 | 3762 | 6750

OUTCOME MEASURES:

1. Primary Outcome: Antibiotic Prescribing Rate at Index Consultation (Immediate or Delayed)
Description: The primary outcome is the percentage of participants who were prescribed antibiotic treatment (both immediate and delayed) at the index consultation as recorded by the treating physician.
Time Frame: This outcome will be registered immediately at the index consultation (immediately after the intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 466 | 817

2. Secondary Outcome: Clinical Recovery During Follow-up
Description: the duration (in days) until reaching full clinical recovery
Time Frame: This outcome will be checked from the diary (via app for parents) from first day after the intervention until day of full clinical recovery (up to maximum 30 days after after the intervention)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
days | 4.6 (3.5) | 4.7 (3.6)

3. Secondary Outcome: Additional Investigations at Index Consultation and/or During Follow-up
Description: the percentage of subjects receiving additional testing (including, but not limited to (X-Ray, blood tests, urine tests) at index consultation (day 0) and/or during follow-up (day 1 to day 30)
Time Frame: This composite outcome will be registered immediately after the intervention and/or checked from the patient health record from the first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 335 | 517

4. Secondary Outcome: Re-consultation During Follow-up
Description: percentage of subjects who re-consulted their physician during follow-up (day 1 to day 30)
Time Frame: This outcome will be checked from the patient health record from first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 770 | 968

5. Secondary Outcome: Antibiotic Prescribing Rate During Follow-up
Description: percentage of subjects who were prescribed antibiotic treatment during follow-up (day 1 to day 30)
Time Frame: This outcome will be checked from the patient health record first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 291 | 429

6. Other Pre Specified Outcome: Additional Testing at Index Consultation
Description: percentage of subjects receiving additional testing (including, but not limited to (X-Ray, blood tests, urine tests) at index consultation (day 0)
Time Frame: This outcome will be registered immediately at the index consultation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 249 | 400

7. Other Pre Specified Outcome: Additional Testing During Follow-up
Description: percentage of subjects receiving additional testing (including, but not limited to (X-Ray, blood tests, urine tests) during follow-up (day 1 to day 30)
Time Frame: during follow-up from first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 111 | 149

8. Other Pre Specified Outcome: Referral to Hospital at Day 0
Description: percentage of subjects referred to hospital at index consultation (day 0)
Time Frame: This outcome will be registered immediately at the index consultation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 24 | 13

9. Other Pre Specified Outcome: Referral to Hospital During Follow-up
Description: percentage of subjects referred to hospital during follow-up (day 1 to day 30)
Time Frame: during follow-up from first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 79 | 84

10. Other Pre Specified Outcome: Admission to Hospital at Day 0
Description: percentage of subjects admitted to hospital at index consultation (day 0)
Time Frame: This outcome will be registered immediately at the index consultation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 7 | 11

11. Other Pre Specified Outcome: Admission to Hospital During Follow-up
Description: percentage of subjects admitted to hospital during follow-up (day 1 to day 30)
Time Frame: during follow-up from first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 25 | 53

12. Other Pre Specified Outcome: Mortality at Day 0
Description: percentage of subjects who died at index consultation (day 0)
Time Frame: This outcome will be registered immediately at the index consultation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 0 | 0

13. Other Pre Specified Outcome: Mortality During Follow up
Description: percentage of subjects who died during follow-up (day 1 to day 30)
Time Frame: during follow-up from first day to day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 0 | 0

14. Other Pre Specified Outcome: Clinical Recovery at Day 7
Description: percentage of subjects with full clinical recovery at day 7
Time Frame: at day 7 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 2539 | 3200

15. Other Pre Specified Outcome: Clinical Recovery at Day 30
Description: percentage of subjects with full clinical recovery at day 30
Time Frame: at day 30 after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
Number analyzed (Participants) | 2988 | 3762
Participants | 2967 | 3747

16. Other Pre Specified Outcome: Patient's Experience Through Semi-structured Interviews
Description: Patient's experience through semi-structured interviews with pre-defined topic guide
Time Frame: within 7 days after the intervention
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Parent's Experience Through Semi-structured Interviews
Description: Parent's experience through semi-structured interviews with pre-defined topic guide
Time Frame: within 7 days after the intervention
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Physician's Experience Through Semi-structured Interviews
Description: Physician's experience through semi-structured interviews with pre-defined topic guide
Time Frame: within 7 days after the intervention
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Cost-effectiveness of the Intervention
Description: Cost-effectiveness of the intervention: healthcare expenditures in terms of hospitalization, consultations, pharmaceuticals (reimbursed and non-reimbursed), productivity, quality of life
Time Frame: will be assessed retrospectively after data collection has finished (24 months of recruitment)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Number of Participants Whose Physician Was Non-Adherent to the Diagnostic Algorithm
Description: clinicians could deviate from the proposed diagnostic algorithm. This outcome measure comprise the percentage of participants whose physician was non-adherent to the diagnostic algorithm. This is not a protocol violation, since deviating from the algorithm was a possibility if the physician deems this necessary.
Time Frame: This outcome will be registered immediately at the index consultation
Population: missing data from 2 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Diagnostic Algorithm
Number analyzed (Participants) | 2986
Participants | 160

ADVERSE EVENTS:
Time Frame: 30 days
Description: Admission to hospital at the index consultation + Admission to hospital day 1-30
Arm/Group | Intervention: Diagnostic Algorithm | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/2988 | 0/3762
Serious Adverse Events (participants affected / at risk) | 0/2988 | 0/3762
Other Adverse Events (participants affected / at risk) | 32/2988 | 64/3762
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Diagnostic Algorithm (N=2988) | Usual Care (N=3762)
hospitalisation (Infections and infestations) | 32 (32) | 64 (64) — hospitalisation due to infections, not caused by the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may only publish the Results provided that Sponsor has duly published the main Study publication. Once the main Study publication has been duly published by the Sponsor, Investigator are entitled to publish the Results provided that Sponsor has granted its prior written approval with Principal Investigator's proposed publication.

DOCUMENTS (3):
  • Study Protocol (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04470518/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT04470518/SAP_001.pdf
  • Informed Consent Form (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT04470518/ICF_002.pdf